CLINICAL TRIAL: NCT00957983
Title: EP4-receptor Antagonism and Prostaglandin E2 (PGE2) in a Human Headache Model
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Messoud Ashina, PhD, dr.med, senior consulter, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BGC20-1531-04
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2009-09

CONDITIONS: Headache, Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — N-(4-(4-(5-methoxypyridin-2-yl)phenoxymethyl)-5-methylfuran-2-carbonyl)-2-methylbenzenesulfonamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- BGC20-1531 200mg (Active Comparator)
  Interventions: Drug: BGC20-1531
- sugar pill (Placebo Comparator)
  Interventions: Drug: BGC20-1531
- BGC20-1531 400mg (Active Comparator)
  Interventions: Drug: BGC20-1531

INTERVENTIONS:
Drug: BGC20-1531 — oral administration followed by Prostaglandin E2 infusion
  Other Names: EP-4 receptor antagonist

SUMMARY:
The purpose of this study is to determine whether EP-4 receptor antagonist can prevent the headache expected during a Prostaglandin E2 infusion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Tension headache
* All other primary forms of headache
* Cardiovascular, Central Nervous system (CNS) and autoimmune diseases
* Gastrointestinal disease
* Previous or clinical signs of mental illness or substance abuse.
* Participation in a clinical study of a medicinal product without regulatory approval or marketing authorisation within 1 month prior to this trial
* Pregnancy/nursing
* Daily intake of medication (except oral contraceptives)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2009-08; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Headache | 24 hours

SECONDARY OUTCOMES:
rCBF, blood flow, diameter of STA/RA, HR, BP | in-hospital

CONTACTS AND LOCATIONS:
Overall Officials: Messoud Ashina, MD, PhD, Principal Investigator — Danish Headache Center
Locations (1):
- Danish Headache Center, Glostrup Municipality, Denmark